CLINICAL TRIAL: NCT06793969
Title: Swartz Sheath With Angioplasty Guidewire-Assisted Versus Conventional Technique for Patent Foramen Ovale Closure: A Multicenter Randomized Controlled Trial
Brief Title: Swartz Sheath With Angioplasty Guidewire-Assisted Technique for Patent Foramen Ovale Closure (STAGE-PFO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STAGE-PFO
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Patent Oval Foramen
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional group (Sham Comparator): In the conventional group, the PFO closure procedure is performed with a multi-functional catheter and guided by intraprocedural fluoroscopy and intracardiac echocardiography (ICE).
  Interventions: Procedure: Conventional technique to pass the PFO tunnel
- The Swartz sheath + angioplasty guidewire group (Active Comparator): In the Swartz sheath + angioplasty guidewire group, the PFO closure procedure is performed with Swartz sheath + angioplasty guidewire assistance and guided by intraprocedural fluoroscopy and ICE.
  Interventions: Procedure: Swartz sheath with Angioplasty Guidewire-Assisted Technique for PFO tunnel passage

INTERVENTIONS:
Procedure: Swartz sheath with Angioplasty Guidewire-Assisted Technique for PFO tunnel passage — The angioplasty guidewire is advanced into the left atrium and left superior pulmonary vein (LSPV). The Swartz sheath is then delivered to the left atrium along the 0.014" guidewire through the PFO. Next, the Runthrough guidewire is changed to a 0.035" J-tipped guidewire, which is advanced into the LSPV. Finally, the delivery sheath for the PFO closure device is introduced to the left atrium along the guidewire, and all other toolkits are withdrawn.
  Arms: The Swartz sheath + angioplasty guidewire group
Procedure: Conventional technique to pass the PFO tunnel — In the conventional group, the PFO closure procedure is performed with a multi-functional catheter and guided by intraprocedural fluoroscopy and ICE
  Arms: The conventional group

SUMMARY:
The technical challenge in patent foramen ovale (PFO) closure lies in successfully establishing an occlusion pathway through the PFO tunnel using a guidewire or catheter. In this study, we aim to investigate the efficacy and safety of Swartz sheath with angioplasty guidewire-assisted technique for PFO Closure.

DETAILED DESCRIPTION:
In cases of complex PFO, failure of guidewire passage through the septum can occur, rendering closure impossible. The present multicenter, prospective, randomized controlled trial aims to evaluate the efficacy and safety of a novel Swartz sheath with angioplasty guidewire-assisted technique to facilitate PFO tunnel passage.

With written consent, the investigators expect to enrol PFO patients with a history of cryptogenic stroke (CS) or transient ischemic attack (TIA), who requires PFO closure according to current guidelines. A standardized TEE protocol is used to assess the morphologic characteristics of the atrial septum and right-to-left shunting through PFO. Eligible patients are prospectively and randomly assigned to the Swartz sheath + angioplasty guidewire group or the conventional group (1:1 ratio). In the Swartz sheath + angioplasty guidewire group, the PFO closure procedure is performed with Swartz sheath + angioplasty guidewire assistance. In the conventional group, the PFO closure procedure is performed with a multi-functional catheter. After the procedure, safety parameters such as contrast use, procedure time, and severe complications are recorded. All patients are followed up at 1-, 3-, 6-, and 12- month post device implantation. The presence of a residual shunt, device embolization, device migration and residual shunt are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65
* Confirmed diagnosis of PFO by transthoracic and transesophageal echocardiography
* A history of cryptogenic stroke (CS) or transient ischemic attack (TIA)

Exclusion Criteria:

* Confirmed pregnancy
* Confirmed diagnosis of intracardiac thrombosis
* Confirmed diagnosis of pulmonary hypertension
* Confirmed diagnosis of rheumatic heart disease, or valvular heart disease
* Past medical history of myocardial infarction, unstable angina and intracranial hemorrhage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-24 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Time of PFO tunnel passage | Intraprocedural assessment (measured in minutes )
  The total time required to pass the guide across PFO tunnel

SECONDARY OUTCOMES:
Procedure Time | Intraprocedural assessment (measured in minutes )
  The total time required to complete PFO closcure
Fluoroscopy Time | Intraprocedural assessment (measured in minutes )
  The total fluoroscopy time during the procedure
Procedural Complications | Intraprocedural assessment
  Complications such as inguinal haematoma and pericardial effusion related to the PFO closure procedure
Radiation Dose | Intraprocedural assessment (measured in mGys)
  The total dosage of radiation required to complete the PFO closure procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China